CLINICAL TRIAL: NCT06498271
Title: Personalized and Automated Digital Coaching in People With Non-specific Chronic Low Back Pain: a Randomized Controlled Trial Nested in the "ComPaRe" E-cohort
Brief Title: Personalized and Automated Digital Coaching in People With Non-specific Chronic Low Back Pain
Acronym: BACK-4P
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Arthritis Foundation (Other); Societe Francaise de Rhumatologie (Other); Association Malakoff Médéric Innovation Santé (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP200223; 2020-A00100-39 (Other: ID-RCB)
Record Dates: First submitted 2024-06-20; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Digital coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Personalized and automated digital coaching smartphone application
  Interventions: Device: Personalized and automated digital coaching using a mobile application
- Comparator group (No Intervention): Usual care

INTERVENTIONS:
Device: Personalized and automated digital coaching using a mobile application — Participants allocated to the experimental group will be invited to download a smartphone application which will appraise their motivation and automatically propose: 1) exercises to be performed at home and adapted to their pain levels; 2) audio recordings for pain management; and 3) educational and coaching content adapted to their motivation. In addition, the smartphone application enables users to plan their home exercises
  Arms: Experimental group

SUMMARY:
The investigators hypothesize that a personalized and automated digital coaching could reduce activity limitations in people with chronic low back pain as compared to usual care

DETAILED DESCRIPTION:
Non-specific low back pain (LBP) is the leading cause of years of life lived with disability worldwide and its burden is growing alongside the increasing and ageing population.

LBP is usually treated according to symptoms duration, presence of concomitant radicular pain and of consistent anatomical abnormalities and is defined according to symptoms duration: acute (< 6 weeks), subacute (6 to 12 weeks) and chronic (> 12 weeks). The prognosis of acute LBP is excellent, but in 5 to 15% of individuals, LBP becomes chronic. At 6 months, about 10% of individuals with chronic LBP are on sick leave, and at 12 months, 20% report persistent disability.

Unfavourable evolution of chronic LBP is characterized by onset and persistence of spine-specific disability in all individuals and work absenteeism in working age individuals. The probability of returning to work is only 20% after 1 year of sick leave and 0% after 2 years. Multidisciplinary rehabilitation that combines education, physical therapy, cognitive behavioural therapy and rehabilitation is usually offered. However, lack of personalization of these programs could affect their efficacy and systematic evaluation suggests their low cost-effectiveness).

Current management of non-specific chronic low back pain involves a multidisciplinary approach that typically includes non-opioid analgesics, physical exercise and strength training, education, and cognitive behavioural therapies. Therapeutic interventions such as massage, acupuncture, or spinal manipulation may also be beneficial.

The investigators hypothesize that a personalized and automated digital coaching could reduce activity limitations in people with chronic LBP, as compared to usual care.

Participants allocated to the experimental group will be invited to download a smartphone application which will appraise their motivation and automatically propose 1) exercises to be performed at home and adapted to their pain levels; 2) audio recordings for pain management; and 3) educational and coaching content adapted to their motivation. In addition, the smartphone application enables users to plan their home exercises.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over
* Having non-specific chronic LBP
* Participating in the "ComPaRe" e-cohort
* Having provided consent for their data to be used to assess trial eligibility

  * And to be randomized if eligible
  * And to, allow their data to be used to evaluate intervention effectiveness without being notified that they are in the control group, if randomized to usual the control group
* Having a valid email address
* Able to read and write French Having a smartphone functioning with Android acquired after 2020

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean change in activity limitations | 4 months
  French version of the self-administered Roland Morris Disability Questionnaires (RMDQ). Higher scores indicate worse function

SECONDARY OUTCOMES:
Mean change in activity limitations at 12 months after consent | 12 months
  French version of the self-administered Roland Morris Disability Questionnaires (RMDQ). Higher scores indicate worse function
Mean change in the intensity of low back pain at 4 months after consent | 4 months
  Self-administered numerical scale with 11 classes incremented by 10 points (0, no pain and 100, maximum pain)
Mean change in the intensity of low back pain at 12 months after consent | 12 months
  Self-administered numerical scale with 11 classes incremented by 10 points (0, no pain and 100, maximum pain)
Work absenteeism at 4 months after consent | 4 months
  Number of self-reported days off work
Work absenteeism at 12 months after consent | 12 months
  Number of self-reported days off work

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, Principal Investigator — Assistance Publique - Hôpitaux de Paris; François RANNOU, MD,PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis - hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ComPaRe ("Communauté de Patients pour la Recherche") is a collaborative open e-cohort of patients with chronic conditions. Within the ComPaRe platform, a cohort specific to non-specific low back pain was launched — https://compare.aphp.fr/lombalgie-chronique/
- See also: click here for more information about this study Back-4P — https://www.back-4p.org/